CLINICAL TRIAL: NCT03428672
Title: Collection of Bone Specimens for Quantitative Analysis of Global Proteome and Iron Content Detection
Brief Title: Quantitative Analysis of Global Proteome in Bone Samples From Patients With Osteoporotic and Nonosteoporotic Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, You-Jia Xu, Director, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Xu youjia 003
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteoporotic fractures (Experimental): patients with osteoporotic fractures, including femoral neck fracture and pertrochanteric fracture. Total hip arthroplasty or proximal femoral nails was needed.
  Interventions: Procedure: total hip arthroplasty
- nonosteoporotic fractures (Sham Comparator): patients with nonosteoporotic fractures, including femoral neck fracture and pertrochanteric fracture. Total hip arthroplasty or proximal femoral nails was needed.
  Interventions: Procedure: total hip arthroplasty

INTERVENTIONS:
Procedure: total hip arthroplasty — Bone samples from Hip fracture were collected from the femoral head which has been replaced

SUMMARY:
RATIONALE: Collecting and storing bone samples from patients with osteoporotic and nonosteoporotic fracture to quantitatively analyze the differentially expressed proteins to further explain the relationship between bone iron content and bone mineral density (BMD).

PURPOSE: This research study is looking at changes of iron content and differentially expressed proteins in bone samples from patients with osteoporotic and nonosteoporotic.

fracture.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Establish the iron content in bone specimen in patients with hip fracture.
2. Explore the correlation of BMD and differentially expressed proteins.

OUTLINE:

1. Collect human bone specimens from patients with osteoporotic and nonosteoporotic Fracture.
2. Provide a repository for storage of tissue and make these specimens available for approved projects by laboratory-based investigators.
3. Collect clinical data on these patients including bone mineral density.
4. To examine the bone iron content using ICP/MS.
5. Investigate the differentially expressed proteins through quantitative analysing the global proteome of osteoporotic and nonosteoporotic fracture bone specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: 55-90 Years
2. Genders Eligible for Study: Woman
3. Accepts Healthy Volunteers: NO
4. Study Population: Female patients with hip fracture.

Exclusion Criteria:

1. Malignancy or benign ovarian cysts
2. Known chronic or systemic diseases
3. Hormone therapy in the previous 3 months
4. Bone metabolism and drug therapy

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
the iron content in human bone samples | 3 month
  Bone samples were preprocess and decomposed by microwave.Icp-ms is used for quantitative detection of samples.

SECONDARY OUTCOMES:
The value of bone mineral density | one week
  Bone mineral density was measured by double energy X-ray absorptiometer (DXA) in a week before surgery.
Quantitative Analysis of Global Proteome in bone samples | 5 month
  Find the differentially expressed proteins in nonosteoporotic or osteoporotic bone sample through using an integrated approach involving TMT labeling and LC-MS/MS to quantify the dynamic changes of the whole proteome of Human Species.

CONTACTS AND LOCATIONS:
Overall Officials: Youjia Xu, PhD, Study Chair — Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiagnsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Geyer PE, Wewer Albrechtsen NJ, Tyanova S, Grassl N, Iepsen EW, Lundgren J, Madsbad S, Holst JJ, Torekov SS, Mann M. Proteomics reveals the effects of sustained weight loss on the human plasma proteome. Mol Syst Biol. 2016 Dec 22;12(12):901. doi: 10.15252/msb.20167357. PMID 28007936
- [Result] Roumeliotis TI, Williams SP, Goncalves E, Alsinet C, Del Castillo Velasco-Herrera M, Aben N, Ghavidel FZ, Michaut M, Schubert M, Price S, Wright JC, Yu L, Yang M, Dienstmann R, Guinney J, Beltrao P, Brazma A, Pardo M, Stegle O, Adams DJ, Wessels L, Saez-Rodriguez J, McDermott U, Choudhary JS. Genomic Determinants of Protein Abundance Variation in Colorectal Cancer Cells. Cell Rep. 2017 Aug 29;20(9):2201-2214. doi: 10.1016/j.celrep.2017.08.010. PMID 28854368
- [Result] Zeng Y, Zhang L, Zhu W, Xu C, He H, Zhou Y, Liu YZ, Tian Q, Zhang JG, Deng FY, Hu HG, Zhang LS, Deng HW. Corrigendum to "Quantitative proteomics and integrative network analysis identified novel genes and pathways related to osteoporosis" [J. Proteomics 142 (16 June 2016) 45-52]. J Proteomics. 2017 Jun 6;162:155. doi: 10.1016/j.jprot.2017.05.023. No abstract available. PMID 28578906
- [Result] Kuo HW, Kuo SM, Chou CH, Lee TC. Determination of 14 elements in Taiwanese bones. Sci Total Environ. 2000 Jun 8;255(1-3):45-54. doi: 10.1016/s0048-9697(00)00448-4. PMID 10898394
- [Result] Brodziak-Dopierala B, Kwapulinski J, Sobczyk K, Wiechula D. The content of manganese and iron in hip joint tissue. J Trace Elem Med Biol. 2013 Jul;27(3):208-12. doi: 10.1016/j.jtemb.2012.12.005. Epub 2013 Feb 15. PMID 23415599